CLINICAL TRIAL: NCT01204398
Title: An Open-label Study to Evaluate the Antihypertensive Effects of the Fixed-dose Combination of Telmisartan 80 mg and Amlodipine 5 mg (T80/A5) Given Once Daily by 24 h ABPM in Patients With Moderate to Severe Hypertension
Brief Title: Telmisartan+Amlodipine Fixed Dose Combination in Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1235.31
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan amlodipine combination

ARMS (1):
- eligible hypertension patient (Experimental): Patients will be given placebo for 2 weeks for wash-out, then qualified patients will be administered Telmisartan 80mg/Amlodipine 5mg for 8 weeks.
  Interventions: Drug: telmisartan+amlodipine fixed dose combination

INTERVENTIONS:
Drug: telmisartan+amlodipine fixed dose combination — after 2 weeks placebo wash-out, patients will be administered Telmisartan 80mg/Amlodipine 5mg for 8 weeks.

SUMMARY:
The primary objectives of this trial is to evaluate the changes from baseline (Visit 2) in the 24-hour Ambulatory Blood Pressure Monitoring mean (relative to dose time) for diastolic blood pressure and systolic blood pressure after 8 weeks of treatment with Telmisartan 80mg/Amlodipine 5mg in patients with moderate to severe hypertension

ELIGIBILITY:
Inclusion criteria:

1. Aged at least 18 years at the date of signing the consent form
2. For treatment-naïve patients: hypertension defined by a mean seated diastolic blood pressure (DBP) equal or more than 100 mmHg measured by manual cuff sphygmomanometry at visit 1 and 2; For pretreatment patients: hypertension defined by a mean seated diastolic blood pressure equal or more than 90 mmHg at visit 1 and equal or more than 100 mmHg at visit 2 measured by manual cuff sphygmomanometry
3. 24-hour mean diastolic blood pressure equal or more than 85 mmHg at baseline Ambulatory Blood Pressure Monitoring

Exclusion criteria:

1. mean seated systolic blood pressure equal or more than 200 mmHg and/or mean seated diastolic blood pressure equal or more than 120 mmHg
2. any clinically significant hepatic impairment
3. severe renal impairment
4. bilateral renal artery stenosis or renal artery stenosis in a solitary kidney or post-renal transplant
5. current treatment with any antihypertensive agents, whether or not prescribed for this indication, that cannot be safely stopped
6. other conditions or situations that could put potential participants at unacceptable risk due to participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1235.31.86001 Boehringer Ingelheim Investigational Site, Shanghai, China

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label study with one treatment arm. Whilst 40 patients were enrolled, 39 entered the placebo run-in and 27 were treated. Therefore the treated set (TS) comprises 27 patients and the full analysis set (FAS) comprises 25 patients.
Groups:
- T80/A5: Telmisartan 80mg plus Amlodipine 5mg fixed-dose combination
Period: Overall Study
Arm/Group | T80/A5
Started | 27 (Entered and treated.)
Completed | 26 (Completed trial medication.)
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | T80/A5
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Mean 24-hour mean Diastolic blood pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 95.79 (7.74)
Mean 24-hour mean Systolic blood pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 150.24 (17.30)

OUTCOME MEASURES:

1. Primary Outcome: DBP and SBP Change From Baseline in Mean 24-hour Ambulatory Blood Pressure Monitoring (ABPM) Mean
Description: ABPM measurements were taken every 20 minutes throughout the day and night by the validated SpaceLabs Model 90217 monitor.
Time Frame: 8 weeks
Population: Full analysis set (FAS) defined as all patients with at least one dose of T80/A5, and for whom baseline and post-baseline ABPM are available.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | T80/A5
Number analyzed (Participants) | 25
mmHg
  DBP change from baseline | -12.76 (7.42)
  SBP change from baseline | -23.82 (14.54)

2. Secondary Outcome: Change From Baseline in ABPM Hourly Mean DBP and SBP, Starting 1 Hour After Dosing
Description: Changes from baseline in DBP and SBP hourly means over the 24-hour dosing interval as measured by ABPM after 8 weeks of treatment with T80/A5
Time Frame: 8 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | T80/A5
Number analyzed (Participants) | 25
mmHg
  DBP Change from baseline after 1 hour | -12.5 (10.7)
  DBP Change from baseline after 2 hours | -14.7 (14.2)
  DBP Change from baseline after 3 hours | -13.7 (13.9)
  DBP Change from baseline after 4 hours | -11.7 (10.9)
  DBP Change from baseline after 5 hours | -9.9 (15.6)
  DBP Change from baseline after 6 hours | -11.7 (13.4)
  DBP Change from baseline after 7 hours | -15.9 (12.3)
  DBP Change from baseline after 8 hours | -14.8 (9.2)
  DBP Change from baseline after 9 hours | -13.7 (11.1)
  DBP Change from baseline after 10 hours | -12.9 (13.3)
  DBP Change from baseline after 11 hours | -13.6 (13.0)
  DBP Change from baseline after 12 hours | -13.1 (12.5)
  DBP Change from baseline after 13 hours | -13.2 (12.4)
  DBP Change from baseline after 14 hours | -11.9 (14.8)
  DBP Change from baseline after 15 hours | -11.5 (12.8)
  DBP Change from baseline after 16 hours | -11.8 (18.3)
  DBP Change from baseline after 17 hours | -12.6 (14.0)
  DBP Change from baseline after 18 hours | -13.1 (12.2)
  DBP Change from baseline after 19 hours | -11.8 (10.6)
  DBP Change from baseline after 20 hours | -10.7 (13.2)
  DBP Change from baseline after 21 hours | -9.0 (13.4)
  DBP Change from baseline after 22 hours | -13.8 (15.8)
  DBP Change from baseline after 23 hours | -13.9 (9.8)
  DBP Change from baseline after 24 hour | -14.8 (12.1)
  SBP Change from baseline after 1 hour | -25.0 (21.3)
  SBP Change from baseline after 2 hours | -26.2 (22.7)
  SBP Change from baseline after 3 hours | -30.1 (26.3)
  SBP Change from baseline after 4 hours | -21.9 (20.3)
  SBP Change from baseline after 5 hours | -23.9 (19.7)
  SBP Change from baseline after 6 hours | -23.9 (22.6)
  SBP Change from baseline after 7 hours | -29.2 (18.8)
  SBP Change from baseline after 8 hours | -27.6 (18.0)
  SBP Change from baseline after 9 hours | -27.7 (21.1)
  SBP Change from baseline after 10 hours | -25.8 (20.2)
  SBP Change from baseline after 11 hours | -22.8 (20.4)
  SBP Change from baseline after 12 hours | -23.4 (19.2)
  SBP Change from baseline after 13 hours | -22.4 (19.5)
  SBP Change from baseline after 14 hours | -22.1 (20.8)
  SBP Change from baseline after 15 hours | -22.9 (19.4)
  SBP Change from baseline after 16 hours | -24.4 (22.5)
  SBP Change from baseline after 17 hours | -23.3 (19.9)
  SBP Change from baseline after 18 hours | -21.7 (22.2)
  SBP Change from baseline after 19 hours | -21.2 (16.8)
  SBP Change from baseline after 20 hours | -20.5 (21.2)
  SBP Change from baseline after 21 hours | -17.0 (24.6)
  SBP Change from baseline after 22 hours | -19.2 (25.8)
  SBP Change from baseline after 23 hours | -24.6 (15.6)
  SBP Change from baseline after 24 hour | -25.1 (16.9)

3. Secondary Outcome: Trough to Peak (T/P) Ratio for DBP and SBP After 8 Weeks of Treatment
Description: Calculated on the basis of changes in hourly means from baseline. Trough is defined as the mean of the last three hours of the 24-hour dosing interval. Peak is the greatest reduction in hourly means in hours 2 to 8 after dosing. All measurements are using ABPM.
Time Frame: 8 weeks
Population: FAS
Measure: Median (Full Range); unit: Ratio
Arm/Group | T80/A5
Number analyzed (Participants) | 25
Ratio
  DBP T/P ratio (N=23) | 1.13 (-14.9, 15.8) [-14.9 to 15.8]
  SBP T/P ratio (N=25) | 0.98 (-7.6, 14.0) [-7.6 to 14.0]

4. Secondary Outcome: Change From Baseline to End of Study in DBP and SBP
Description: Manually measured in-clinic DBP and SBP
Time Frame: 8 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | T80/A5
Number analyzed (Participants) | 25
mmHg
  DBP: Change from baseline to 2 weeks | -9.67 (7.14)
  DBP: Change from baseline to 4 weeks | -13.49 (7.22)
  DBP: Change from baseline to 8 weeks | -13.73 (6.58)
  SBP: Change from baseline to 2 weeks | -11.04 (8.99)
  SBP: Change from baseline to 4 weeks | -17.95 (10.53)
  SBP: Change from baseline to 8 weeks | -19.80 (9.96)

5. Secondary Outcome: ABPM Hourly Mean DBP and SBP at Baseline and the End of the Study, Starting 1 Hour After Dosing
Description: DBP and SBP hourly means over the 24-hour dosing interval as measured by ABPM at baseline and after 8 weeks of treatment
Time Frame: 0 and 8 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | T80/A5
Number analyzed (Participants) | 25
mmHg
  DBP after 1 hour at baseline | 101.6 (10.2)
  DBP after 2 hours at baseline | 101.7 (13.2)
  DBP after 3 hours at baseline | 100.0 (11.1)
  DBP after 4 hours at baseline | 97.9 (9.5)
  DBP after 5 hours at baseline | 95.3 (11.3)
  DBP after 6 hours at baseline | 96.5 (11.6)
  DBP after 7 hours at baseline | 97.0 (12.6)
  DBP after 8 hours at baseline | 100.6 (9.8)
  DBP after 9 hours at baseline | 102.7 (10.3)
  DBP after 10 hours at baseline | 100.4 (11.2)
  DBP after 11 hours at baseline | 97.9 (11.8)
  DBP after 12 hours at baseline | 95.9 (11.0)
  DBP after 13 hours at baseline | 93.6 (11.8)
  DBP after 14 hours at baseline | 92.0 (11.5)
  DBP after 15 hours at baseline | 89.4 (11.9)
  DBP after 16 hours at baseline | 89.1 (16.8)
  DBP after 17 hours at baseline | 88.0 (10.4)
  DBP after 18 hours at baseline | 88.8 (11.6)
  DBP after 19 hours at baseline | 88.4 (10.3)
  DBP after 20 hours at baseline | 90.3 (12.9)
  DBP after 21 hours at baseline | 91.4 (10.4)
  DBP after 22 hours at baseline | 97.6 (14.2)
  DBP after 23 hours at baseline | 101.0 (10.0)
  DBP after 24 hours at baseline | 101.8 (9.3)
  DBP after 1 hour at the end of the study | 89.1 (8.5)
  DBP after 2 hours at the end of the study | 87.1 (11.0)
  DBP after 3 hours at the end of the study | 86.3 (11.1)
  DBP after 4 hours at the end of the study | 86.2 (10.1)
  DBP after 5 hours at the end of the study | 85.3 (10.2)
  DBP after 6 hours at the end of the study | 84.8 (11.4)
  DBP after 7 hours at the end of the study | 81.1 (12.8)
  DBP after 8 hours at the end of the study | 85.8 (7.5)
  DBP after 9 hours at the end of the study | 88.9 (9.7)
  DBP after 10 hours at the end of the study | 87.5 (10.5)
  DBP after 11 hours at the end of the study | 84.3 (9.6)
  DBP after 12 hours at the end of the study | 82.8 (9.1)
  DBP after 13 hours at the end of the study | 80.4 (10.2)
  DBP after 14 hours at the end of the study | 80.1 (13.6)
  DBP after 15 hours at the end of the study | 77.9 (11.4)
  DBP after 16 hours at the end of the study | 77.3 (8.9)
  DBP after 17 hours at the end of the study | 75.5 (11.2)
  DBP after 18 hours at the end of the study | 75.7 (11.5)
  DBP after 19 hours at the end of the study | 76.6 (9.7)
  DBP after 20 hours at the end of the study | 79.6 (10.4)
  DBP after 21 hours at the end of the study | 82.4 (10.5)
  DBP after 22 hours at the end of the study | 83.8 (12.5)
  DBP after 23 hours at the end of the study | 87.2 (10.4)
  DBP after 24 hours at the end of the study | 87.0 (12.4)
  SBP after 1 hour at baseline | 157.9 (17.9)
  SBP after 2 hours at baseline | 156.5 (20.1)
  SBP after 3 hours at baseline | 158.4 (21.4)
  SBP after 4 hours at baseline | 152.6 (15.9)
  SBP after 5 hours at baseline | 152.1 (21.1)
  SBP after 6 hours at baseline | 152.6 (24.6)
  SBP after 7 hours at baseline | 154.6 (23.3)
  SBP after 8 hours at baseline | 157.3 (19.6)
  SBP after 9 hours at baseline | 161.0 (18.6)
  SBP after 10 hours at baseline | 157.6 (20.2)
  SBP after 11 hours at baseline | 153.3 (21.8)
  SBP after 12 hours at baseline | 150.0 (20.8)
  SBP after 13 hours at baseline | 145.8 (22.2)
  SBP after 14 hours at baseline | 146.3 (22.7)
  SBP after 15 hours at baseline | 141.9 (23.9)
  SBP after 16 hours at baseline | 142.2 (26.2)
  SBP after 17 hours at baseline | 139.6 (19.1)
  SBP after 18 hours at baseline | 137.8 (22.9)
  SBP after 19 hours at baseline | 139.2 (20.5)
  SBP after 20 hours at baseline | 142.2 (21.6)
  SBP after 21 hours at baseline | 143.6 (20.6)
  SBP after 22 hours at baseline | 148.5 (22.2)
  SBP after 23 hours at baseline | 156.6 (18.9)
  SBP after 24 hours at baseline | 158.2 (16.6)
  SBP after 1 hour at the end of the study | 132.8 (15.0)
  SBP after 2 hours at the end of the study | 130.2 (15.3)
  SBP after 3 hours at the end of the study | 128.3 (17.9)
  SBP after 4 hours at the end of the study | 130.6 (17.8)
  SBP after 5 hours at the end of the study | 128.2 (19.1)
  SBP after 6 hours at the end of the study | 128.8 (17.3)
  SBP after 7 hours at the end of the study | 125.5 (19.4)
  SBP after 8 hours at the end of the study | 129.7 (15.5)
  SBP after 9 hours at the end of the study | 133.2 (16.8)
  SBP after 10 hours at the end of the study | 131.7 (17.3)
  SBP after 11 hours at the end of the study | 130.5 (17.8)
  SBP after 12 hours at the end of the study | 126.6 (15.9)
  SBP after 13 hours at the end of the study | 123.5 (15.8)
  SBP after 14 hours at the end of the study | 124.2 (19.9)
  SBP after 15 hours at the end of the study | 119.1 (14.6)
  SBP after 16 hours at the end of the study | 117.8 (14.6)
  SBP after 17 hours at the end of the study | 116.4 (16.0)
  SBP after 18 hours at the end of the study | 116.1 (18.4)
  SBP after 19 hours at the end of the study | 118.0 (17.8)
  SBP after 20 hours at the end of the study | 121.7 (19.0)
  SBP after 21 hours at the end of the study | 126.6 (18.3)
  SBP after 22 hours at the end of the study | 129.3 (21.5)
  SBP after 23 hours at the end of the study | 132.0 (16.6)
  SBP after 24 hours at the end of the study | 133.1 (20.2)

6. Secondary Outcome: Treatment Emergent Adverse Events
Description: Electrocardiogram, laboratory parameters and physical examinations were performed and any abnormal findings were recorded within the adverse events
Time Frame: 8 weeks
Population: Treated Set (TS) defined as all patients who entered the run-in phase and were treated with T80/A5.
Measure: Number; unit: Participants
Arm/Group | T80/A5
Number analyzed (Participants) | 27
Participants
  Patients with any AEs | 4
  Patients with severe AEs | 0
  Patients with drug-related AEs | 1
  Patients with AEs related to laboratory changes | 0

7. Secondary Outcome: Change From Baseline to End of Study in In-clinic Pulse Rate
Time Frame: 8 weeks
Population: TS with non-missing data
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | T80/A5
Number analyzed (Participants) | 27
beats per minute (bpm) | 2.37 (5.95)

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- T80/A5: Telmisartan 80 mg plus Amlodipine 5 mg once daily
Arm/Group | T80/A5
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.